CLINICAL TRIAL: NCT06367036
Title: Effect of Hypericum Perforatum Oil on Prevention Ecchymosis and Pain Associated With Subcutaneous Low Molecular Weight Heparin Injection: a Self-controlled Single-blind Study
Brief Title: Effect of Hypericum Perforatum Oil on Ecchymosis and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, HATİCE DEMİRDAĞ, Assistant Proffessor, Uskudar University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-52
Record Dates: First submitted 2024-04-06; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pain; Ecchymosis
Keywords: Hypericum Perforatum oil; low molecular weight heparin; subcutaneous injection; ecchymosis; pain
MeSH Terms: conditions — Pain; Ecchymosis

STUDY DESIGN:
Intervention Model Description: There is no control group in this research design. The participants themselves are also the control group. Intervention was applied to one injection site of the participants 2 hours before the injection and not to the other. Post-injection pain and ecchymosis were evaluated for both sites. The two researchers who analyzed the results do not know the region where the intervention was applied.
Who Masked: Investigator
Masking Description: Two researchers do not know which site was injected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypericum Perforatum Oil group (Experimental): This research is a self-controlled study. One injected arm of the patient will be assigned to the intervention group and the other arm to the control group. İn the experimental arm, the research nurse working in the Coronary Intensive Care unit (CICU) applied 5-6 drops of HP oil on one arm of the patient with a patting motion 2 hours before the injection. The area was left open for the oil to be absorbed. Only this nurse who administered the injection knows on which arm the oil was applied. The assessment of ecchymosis and pain at the injection site was performed by two other investigators at the 48th hour of the injection (Single blind).
  Interventions: Other: Topical hypericum perforatum oil intervention
- Control group (No Intervention): This research is a self-controlled study. One injected arm of the patient will be assigned to the intervention group and the other arm to the control group.In the control arm, no treatment was performed before injection.The assessment of ecchymosis and pain at the injection site was performed by two other investigators at the 48th hour of the injection (Single blind).

INTERVENTIONS:
Other: Topical hypericum perforatum oil intervention — The research nurse working in the CICU applied 5-6 drops of hypericum perforatum oil on one arm of the patient with a patting motion 2 hours before the injection. The area was left open for the oil to be absorbed. Only this nurse who administered the injection knows on which arm the oil was applied.
  Arms: Hypericum Perforatum Oil group

SUMMARY:
Low molecular weight heparin is a drug with anticoagulant and antithrombotic effects. This drug is frequently administered subcutaneously to patients by nurses. Complications such as pain, ecchymosis and hematoma may commonly occur at the injection site. This study investigated the effect of Hypericum Perforatum oil in preventing pain and ecchymosis after subcutaneous injection low molecular weight heparin. This quasi-experimental and single blinded study was conducted with 160 patients in a coronary intensive care unit. The researcher nurse applied 5-6 drops of Hypericum Perforatum oil to one arm of the patients 2 hours before the injection. The other arm of the patient was considered as the control arm. A total of 320 injections were administered. The evaluation of the injection sites was performed by two other researchers at 48th hours. The data were analyzed using Wilcoxon and McNemar test.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Normal platelet value,
* Normal international normalised ratio (INR) and prothrombin time (PTZ) values,
* No infection, scar tissue or incision in the lateral upper arm

Exclusion Criteria:

* Pregnancy
* Administration of haemodialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Pain point | 48 hours after injection
  The patient's pain was evaluated with Visual Analogue Scale (VAS) 48 hours after the injection. Visual Analogue Scale is a reliable pain assessment scale to determine the pain felt by patients at the injection site. The VAS is a self-report scale consisting of a horizontal line (10 cm long) with anchor points "no pain" and "worst possible pain". The patient is asked to mark the place on this line that best describes the intensity of pain. A marking of "0" means "no pain". Marking "10" means "'intolerable pain". In this way, the patient scores his/her pain between 1-10.
Ecchymosis | 48 hours after injection
  Ecchymosis was evaluated at 48th hours after injection in the study. A transparent ruler that allows millimetric measurement was used to measure the ecchymosis at the injection site. The discoloration at the injection site was measured in millimeter. Ecchymosis was defined as an area of discolored skin of more than 2 mm appearing 48th hours after administration. The maximum horizontal extent (diameter) of the bruise was recorded regardless of whether the bruise was regular or uneven in shape at the time of measurement. According to previous studies, bruise size was analyzed according to 3 categories: no bruise (0-1 mm), small bruise (2-5 mm) and large bruise (>5 mm). In our study, bruises >2 mm in size was accepted as ecchymosis.

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan UYSAL, Associate Professor, Study Chair — Üsküdar University; Zehra KAMBER, Study Chair — Siyami Ersek Thoracic and Cardiovascular Surgery Education Research Hospital
Locations (1):
- Hatice Demirdağ, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared if necessary and requested.